CLINICAL TRIAL: NCT01186029
Title: A Comparison Study to Determine the Increased Efficacy of Adding EMEND to the Treatment Regimen for Post-Discharge and Post-Operative Nausea and Vomiting
Brief Title: Comparison of Adding EMEND to PONV/PDNV Treatment Regimen
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It didn't get IRB approval.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0359-09-FB
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMEND Added to the Treatment Regimen for Post-Discharge and Post-Operative Nausea and Vomiting (Active Comparator): The addition of Aprepitant (Emend), an antiemetic, to 2 drugs that are already used as a standard of care for post-operative nausea and vomiting and post-discharge nausea and vomiting.
  Interventions: Drug: aprepitant
- Standard Treatment Regimen for Post-Discharge and Post-Operative Nausea and Vomiting (No Intervention): No addition of Aprepitant (Emend), an antiemetic, to 2 drugs that are already used as a standard of care for post-operative nausea and vomiting and post-discharge nausea and vomiting.

INTERVENTIONS:
Drug: aprepitant — Emend 40mg by mouth 30 minutes before procedure x 1
  Other Names: EMEND
  Arms: EMEND Added to the Treatment Regimen for Post-Discharge and Post-Operative Nausea and Vomiting

SUMMARY:
This study is looking at whether the addition of Aprepitant (Emend), an antiemetic, will provide added efficacy if added to 2 drugs that are already used as a standard of care for post-operative nausea and vomiting and post-discharge nausea and vomiting.

DETAILED DESCRIPTION:
This study is looking at whether the addition of a fairly new drug for the treatment of post-operative nausea and vomiting (PONV) and post-discharge nausea and vomiting (PDNV) will provide added efficacy if added to 2 drugs that are already used as a standard of care for PONV and PDNV.

The patients that will be looked at will be deemed at higher risk for PONV and PDNV based on the procedure they are having done and/or on patient risk factors.

ELIGIBILITY:
Inclusion Criteria:

* patients with at least 2 of the common risk factors for PONV/PDNV; patients having a procedure deemed at high risk for PONV/PDNV

Exclusion Criteria:

* patients under 19 years of age; pregnant and breast-feeding patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-01 (Actual)

PRIMARY OUTCOMES:
EMEND Added to Standard Treatment of Post-operative and Post-Discharge Nausea and Vomiting | 1 year
  To see if by adding EMEND to a standard treatment regimen for PONV/PDNV, added efficacy will be obtained. To see if there is more efficacy for PONV vs. PDNV by adding EMEND to the treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Michaelis, MD, Principal Investigator — University of Nebraska